CLINICAL TRIAL: NCT02151994
Title: A Double-blind, Randomised, Placebo-controlled, Combined Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetic, Including Food Interaction, and Pharmacodynamic Profile of BIA 5-1058, in Healthy Male Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetic, Including Food Interaction, and Pharmacodynamic Profile of BIA 5-1058.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-51058-101
Record Dates: First submitted 2014-05-26; First posted 2014-06-02 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension and Chronic Heart Failure
Keywords: BIA 5-1058; hypertension; chronic heart failure; cardiovascular disorders
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — zamicastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIA 5-1058 (Experimental): BIA 5-1058 (5, 25 and 100 mg) tablets
  Interventions: Drug: BIA 5-1058
- Placebo (Placebo Comparator): tablets, visually matching active medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 5-1058 — oral administration
  Other Names: Zamicastat
  Arms: BIA 5-1058
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to to assess the safety and tolerability of BIA 5 1058 after single and multiple oral doses

DETAILED DESCRIPTION:
This was a Phase 1, double blind, randomised, placebo-controlled combined single ascending dose (SAD), including food interaction (food effect, FE) analysis, and multiple ascending dose (MAD) study.

SAD: This part consisted of an eligibility screening period, one study period involving administration of single doses of BIA 5-1058 or placebo according to a randomized design, and a follow-up period. Nine sequential groups of 8 healthy young male subjects were dosed. Within each group, 6 subjects were randomised to receive BIA 5-1058 and 2 subjects were randomised to receive placebo. In this first-in-human study, the subjects participating at the lowest dose level of 5 mg were dosed according to a sentinel dosing design to ensure optimal safety. Initially, 2 subjects were dosed; 1 subject with BIA 5-1058 and 1 subject with placebo. After the safety and tolerability results of the first 24 h following dosing for the initial subjects had been found to be acceptable to the MI, the other 6 subjects of the lowest dose level were dosed.

MAD: This part consisted of an eligibility screening period, one study period involving administration of multiple doses of BIA 5-1058 or placebo once daily for 10 days, and a follow-up period. Five sequential groups of 8 healthy young male subjects were dosed.

Within each group, 6 subjects were randomised to receive BIA 5-1058 and 2 subjects were randomised to receive placebo.

The starting dose of 50 mg was chosen taking into consideration the dose range of the previous SAD sequential groups and was approved by the IEC. Escalation to the next higher dose and the determination of the next dose level was based on safety, tolerability and available PK results of the previously administered dose

FE: This part consisted of an eligibility screening period, an open-label two-way crossover study period, and a follow-up period. One group of 12 subjects received single doses of 400 mg BIA 5-1058 during 2 treatment periods, once after having fasted overnight and once after consumption of a high fat breakfast. Each treatment was separated by a period of at least 7 days. The treatment sequence was determined by randomisation.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for the study if they met all the following inclusion criteria:

* Gender - male
* Age - 18 - 55 years, inclusive
* Body Mass Index (BMI) - 18.0 - 30.0 kg m2 (BMI (kg m2) = Body weight (kg) - Heigh t2 (m 2))
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, power drinks), grapefruit (juice) and tobacco products from 48 h prior to entry in the clinical research centre until discharge
* Medical history without major pathology
* Normal resting supine blood pressure and pulse rate showing no clinically relevant deviations as judged by the MI
* Computerised (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the MI
* All values for haematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the MI
* Willingness to sign the written ICF

Exclusion Criteria:

Subjects were excluded from participation if any of the following exclusion criteria applied

* Any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, haematological, neurologic, or psychiatric disease
* An automatic ECG QTc interval reading at screening or enrolment of + 440 ms.
* Evidence of clinically relevant pathology
* Mental handicap
* History of relevant drug and or food allergies
* Smoking more than 10 cigarettes and or cigars and or pipes daily
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
* Use of any prescription drug within 30 days before study drug administration with the exception of influenza vaccination
* Use of any over-the-counter drugs including health supplements, herbal supplements such as St. John's Wort extract (except for the occasional use of acetaminophen (paracetamol), aspirin and vitamins - 100 recommended daily allowance) within 7 days before study drug administration. The use of paracetamol and or topical medication was allowed up to 3 days before entrance into the clinical research facility
* Participation in a drug study within 90 days prior to drug administration
* Participation in more than 3 other drug studies in the 10 months preceding the start of this study (this was the first administration of study drug)
* Donation of more than 50 mL of blood within 90 days prior to first drug administration
* Donation of more than 1.5 litres of blood in the 10 months preceding the start of this study (this was the first administration of study drug)
* Positive screen on drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids), barbiturates, benzodiazepines, tricyclic antidepressants and alcohol
* Intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
* Positive screen on hepatitis B surface antigen (HBsAg)
* Positive screen on anti hepatitis C virus (HCV)
* Positive screen on anti human immunodeficiency virus (HIV) 1 - 2
* Acute disease state indicated as clinically relevant by the MI (e.g. nausea, vomiting, fever, diarrhoea) within 7 days before the first drug administration
* Non-willingness to consume the Food and Drug Administration (FDA) breakfast (FE part only)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA, Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period : Date of first screening to last follow-up: 03 March 2011 - 13 January 2012;
Groups:
- Placebo: Placebo : visually matching active medication
- 5 mg; 25 mg; 800 mg; 1600 mg; 2400 mg: BIA 5-1058 (5, 25 and 100 mg) tablets SAD part: Single dose of BIA 5-1058 (n=6) or matching placebo (n=2) on Day 1, at the following dose levels: 5, 25, 50, 100, 200, 400, 800, 1600 and 2400 mg. Escalation to the next higher dose and any dose adjustments of the next dose levels were based on safety and tolerability results of the previously administered dose and available PK data of previous dose groups.
- 50 mg; 100 mg; 200 mg; 400 mg: BIA 5-1058 (5, 25 and 100 mg) tablets SAD part: Single dose of BIA 5-1058 (n=6) or matching placebo (n=2) on Day 1, at the following dose levels: 5, 25, 50, 100, 200, 400, 800, 1600 and 2400 mg. Escalation to the next higher dose and any dose adjustments of the next dose levels were based on safety and tolerability results of the previously administered dose and available PK data of previous dose groups.
  MAD part: Multiple doses of BIA 5-1058 (n=6) or matching placebo (n=2) once daily on Days 1 to 10, at the following dose levels: 50, 100, 200, 400 and 1200 mg.
- 1200 mg: BIA 5-1058 (5, 25 and 100 mg) tablets MAD part: Multiple doses of BIA 5-1058 (n=6) or matching placebo (n=2) once daily on Days 1 to 10, at the following dose levels: 50, 100, 200, 400 and 1200 mg.
- 400 mg Fasted; 400 mg Fed: BIA 5-1058 (5, 25 and 100 mg) tablets FE part: A single dose of 400 mg BIA 5-1058 on Day 1 under fasted (one period) and fed (one period) conditions.
Period: Single Ascending Dose (SAD)
Arm/Group | Placebo | 5 mg | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg | 800 mg | 1200 mg | 1600 mg | 2400 mg | 400 mg Fasted | 400 mg Fed
Started | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 0 | 0
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Multiple Ascending Dose (MAD)
Arm/Group | Placebo | 5 mg | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg | 800 mg | 1200 mg | 1600 mg | 2400 mg | 400 mg Fasted | 400 mg Fed
Started | 10 | 0 | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 0 | 0
Completed | 10 | 0 | 0 | 6 | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Food Effect (FE): Fasted
Arm/Group | Placebo | 5 mg | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg | 800 mg | 1200 mg | 1600 mg | 2400 mg | 400 mg Fasted | 400 mg Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Food Effect (FE): Fed
Arm/Group | Placebo | 5 mg | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg | 800 mg | 1200 mg | 1600 mg | 2400 mg | 400 mg Fasted | 400 mg Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Ascending Dose (SAD): This part consisted of an eligibility screening period, one study period involving administration of single doses of BIA 5-1058 or placebo according to a randomised design, and a follow-up period. Nine sequential groups of 8 healthy young male subjects were dosed. Within each group, 6 subjects were randomised to receive BIA 5-1058 and 2 subjects were randomised to receive placebo.
- Multiple Ascending Dose (MAD): This part consisted of an eligibility screening period, one study period involving administration of multiple doses of BIA 5-1058 or placebo once daily for 10 days, and a follow-up period. Five sequential groups of 8 healthy young male subjects were dosed. Within each group, 6 subjects were randomised to receive BIA 5-1058 and 2 subjects were randomised to receive placebo.
- Food Interaction (Food Effect, FE) Analysis: This part consisted of an eligibility screening period, an open-label two-way crossover study period, and a follow-up period. One group of 12 subjects received single doses of 400 mg BIA 5-1058 during 2 treatment periods, once after having fasted overnight and once after consumption of a high fat breakfast. Each treatment was separated by a period of at least 7 days. The treatment sequence was determined by randomisation.
- Total: Total of all reporting groups
Arm/Group | Single Ascending Dose (SAD) | Multiple Ascending Dose (MAD) | Food Interaction (Food Effect, FE) Analysis | Total
Number analyzed (Participants) | 72 | 40 | 12 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 0 | 2
  Between 18 and 65 years | 72 | 38 | 12 | 122
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 72 | 40 | 12 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects With Treatment-Emergent Adverse Event (TEAE) Related to Study Medication (SM) - Single Ascending Dose (SAD) Period
Description: Just before drug administration and twice daily until 72 h after (last) drug administration, subjects were asked non-leading questions to determine the occurrence of AEs. Subjects were asked in general terms about any AEs at regular intervals during each study period. In addition, all AEs reported spontaneously during the course of the study were recorded. All answers were assessed by the Medical Investigator (MI), coded using the Medical Dictionary for Regulatory Activities (MedDRA; Version 14.0) and recorded in the AEs Record. The intensity of the AEs was rated as "mild", "moderate" or "severe" and the relationship between the AEs and the study medication was indicated as "not related", "unlikely", "possible", "probable" or ''definite".
Time Frame: Just before drug administration and twice daily until 72 h after (last) drug administration
Measure: Number; unit: % of subject with TEAEs related to SM
Groups:
- 5 mg; 25 mg; 50 mg; 100 mg; 200 mg; 400 mg; 800 mg; 1600 mg; 2400 mg: BIA 5-1058 (5, 25 and 100 mg) tablets
Arm/Group | Placebo | 5 mg | 25 mg | 50 mg | 100 mg | 200 mg | 400 mg | 800 mg | 1600 mg | 2400 mg
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
% of subject with TEAEs related to SM | 28 | 0 | 0 | 0 | 0 | 0 | 17 | 17 | 0 | 67

2. Primary Outcome: Percentage (%) of Subjects With Treatment-Emergent Adverse Event (TEAE) Related to Study Medication (SM) - Multiple Ascending Dose (MAD) Period
Description: as for outcome 1
Time Frame: Just before drug administration and twice daily until 72 h after (last) drug administration
Population: No drug-related TEAEs were reported for the dose levels of 50 mg md and 400 mg md.
Measure: Number; unit: % of subject with TEAEs related to SM
Groups:
- 1200 mg: BIA 5-1058 (5, 25 and 100 mg) tablets
Arm/Group | Placebo | 50 mg | 100 mg | 200 mg | 400 mg | 1200 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
% of subject with TEAEs related to SM | 30 | 0 | 50 | 33 | 0 | 33

3. Primary Outcome: Percentage (%) of Subjects With Treatment-Emergent Adverse Event (TEAE) Related to Study Medication (SM) - Food Effect (FE)
Description: as for outcome 1
Time Frame: Just before drug administration and twice daily until 72 h after (last) drug administration
Measure: Number; unit: % of subject with TEAEs related to SM
Groups:
- 400 mg Fasted; 400 mg Fed: BIA 5-1058 (5, 25 and 100 mg) tablets
Arm/Group | 400 mg Fasted | 400 mg Fed
Number analyzed (Participants) | 12 | 12
% of subject with TEAEs related to SM | 0 | 17

ADVERSE EVENTS:
Time Frame: Just before drug administration and twice daily until 72 h after (last) drug administration
Groups:
- Placebo (SAD); 5 mg (SAD); 25 mg (SAD); 50 mg (SAD); 100 mg (SAD); 200 mg (SAD); 400 mg (SAD); 800 mg (SAD); 1600 mg (SAD); 2400 mg (SAD): SAD period
- 400 mg Fasted (FE Period); 400 mg Fed (FE Period): FE period
- Placebo (MAD Period); 50 mg (MAD Period); 100 mg (MAD Period); 200 mg (MAD Period); 400 mg (MAD Period); 1200 mg (MAD Period): MAD period
Arm/Group | Placebo (SAD) | 5 mg (SAD) | 25 mg (SAD) | 50 mg (SAD) | 100 mg (SAD) | 200 mg (SAD) | 400 mg (SAD) | 800 mg (SAD) | 1600 mg (SAD) | 2400 mg (SAD) | 400 mg Fasted (FE Period) | 400 mg Fed (FE Period) | Placebo (MAD Period) | 50 mg (MAD Period) | 100 mg (MAD Period) | 200 mg (MAD Period) | 400 mg (MAD Period) | 1200 mg (MAD Period)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 11/18 | 0/6 | 2/6 | 3/6 | 2/6 | 4/6 | 4/6 | 3/6 | 1/6 | 4/6 | 3/12 | 5/12 | 8/10 | 5/6 | 3/6 | 5/6 | 3/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SAD) (N=18) | 5 mg (SAD) (N=6) | 25 mg (SAD) (N=6) | 50 mg (SAD) (N=6) | 100 mg (SAD) (N=6) | 200 mg (SAD) (N=6) | 400 mg (SAD) (N=6) | 800 mg (SAD) (N=6) | 1600 mg (SAD) (N=6) | 2400 mg (SAD) (N=6) | 400 mg Fasted (FE Period) (N=12) | 400 mg Fed (FE Period) (N=12) | Placebo (MAD Period) (N=10) | 50 mg (MAD Period) (N=6) | 100 mg (MAD Period) (N=6) | 200 mg (MAD Period) (N=6) | 400 mg (MAD Period) (N=6) | 1200 mg (MAD Period) (N=6)
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
application site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
application site rash (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
catheter site related reaction (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 0 | 0
feeling of relaxation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
headache (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 5
somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
catheter site related inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
feeling drunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other